CLINICAL TRIAL: NCT02986763
Title: Evaluation of Pesticide Exposure in the General Population: Use of Spatial, Environmental, Toxicological and Biological Approaches
Brief Title: Evaluation of Pesticide Exposure in the General Population
Acronym: SIGEXPOSOME
Status: Completed | Type: Observational
Sponsor: Centre Leon Berard (Other)
Collaborators: Cancéropôle Lyon Auvergne Rhône-Alpes (Other); International Agency for Research on Cancer (Other); Rovaltain Research Company (Unknown); Centre de rechercher en Cancérologie de Lyon (Unknown)
Responsible Party: Sponsor
Other Study IDs: SIGEXPOSOME
Record Dates: First submitted 2016-11-30; First posted 2016-12-08 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Pesticide Poisoning
MeSH Terms: interventions — Surveys and Questionnaires; Blood Specimen Collection; Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Professional pesticides: A specific questionnaire with professional information about pesticide uses is added for this arm Questionnaire to collect domestic pesticide use, diet, household characteristics Dust sampling Blood sampling Urine sampling Hair sampling
  Interventions: Biological: Questionnaire, blood, urine, hair and dust samplings
- Volunteers: Questionnaire to collect domestic pesticide use, diet, household characteristics Dust sampling Blood sampling Urine sampling Hair sampling
  Interventions: Biological: Questionnaire, blood, urine, hair and dust samplings

INTERVENTIONS:
Biological: Questionnaire, blood, urine, hair and dust samplings

SUMMARY:
An association has been suggested with several diseases including cancer and IARC has classified several pesticides as carcinogenic, probably carcinogenic. There is a need for a better characterisation of environmental pesticides exposures and identification of suitable biomarkers of exposure and effect. A better understanding of the impact of pesticide exposure on metabolomic, transcriptomic and epigenetic changes, is essential to strengthen epidemiological hypotheses on the association with several cancer types.

The main objective of the project is to validate a GIS (geographic information system) based method to assess environmental pesticide exposures, using environmental (contamination of housedust) and biological (blood and urine samples) measures. The project aims further to investigate a potential link between housedust contamination and biological measures in healthy non-smoking male residents and explore the impact of environmental pesticide exposure on metabolomics, transcriptomic and epigenetic parameters.

DETAILED DESCRIPTION:
The project involves a pilot phase involving repeated (twice) sampling in 20 male non-smoking volunteers living in the Beaujolais region (France) to perform appropriate calibrations for metabolomic, transcriptomic and epigenetic analyses. The main study will be conducted in a sample of 150 male non-smoking volunteers and 50 professional pesticides applicators from the same region (3 sampling periods).

ELIGIBILITY:
Inclusion Criteria:

* Non smokers in the last two years Living in the Beaujolais region (France) within 1000m of vignards Informed consent signed

Exclusion Criteria:

* Volunteers sharing the same households with professional applicators of pesticides

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers living in the Beaujolais region (France)
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2015-06; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
level of pesticide exposures | up to 2 years
  environmental, occupational and domestic exposures